CLINICAL TRIAL: NCT06668415
Title: Effects of Spencer Technique Following Hydrodilation in Patients With Adhesive Capsulitis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Foundation University Islamabad (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FUI/CTR/2024/47
Record Dates: First submitted 2024-10-30; First posted 2024-10-31 (Actual); Last update posted 2024-10-31 (Actual); Status verified 2024-10

CONDITIONS: Adhesive Capsulitis
Keywords: Hydrodilation, spencer technique, pain, functional disability, range of motion
MeSH Terms: conditions — Bursitis; Pain | interventions — Muscle Stretching Exercises

STUDY DESIGN:
Intervention Model Description: This is a randomized controlled trial having two groups. Both groups; Group A and B will undergo Hydrodilation but Group A will be followed by Spencer Technique whereas Group B will be followed by Passive Stretching.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Hydrodilation+Spencer Technique ) (Active Comparator): Patients in this group will be followed by Spencer Technique after Hydrodilation for the duration of 4 weeks which includes 12 sessions in total. Spencer muscle energy technique is a seven 7 step procedure which consists of shoulder extension with elbow flexed, shoulder flexion with elbow flexed, circumduction with compression, circumduction with traction, Abduction then adduction with external rotation and glenohumeral pump. Following the complete action, patients will be encouraged to use their muscles for 3 to 5 seconds against little resistance provided by the therapist
  Interventions: Procedure: Hydro dilation; Procedure: Spencer muscle energy technique
- Group B (Hydro dilation+ Passive Stretching) (Experimental): This group will undergo Passive Stretching followed by Hydrodilation. The low intensity stretches will be given in supine for all the movements ie Flexion ,Abduction , Internal Rotation and External Rotation for 5 repititions with 30 sec hold. (7)
  Interventions: Procedure: Hydro dilation; Procedure: Passive Stretching

INTERVENTIONS:
Procedure: Hydro dilation — The hydro dilation injections comprises of Depomedrol 80mg and normal saline 0.9%. It is performed under fluoroscopic guidance by the orthopedic surgeon.
Procedure: Spencer muscle energy technique — Spencer muscle energy technique is a seven 7 step procedure which consists of shoulder extension with elbow flexed, shoulder flexion with elbow flexed, circumduction with compression, circumduction with traction, Abduction then adduction with external rotation and glenohumeral pump. Following the complete action, patients will be encouraged to use their muscles for 3 to 5 seconds against little resistance provided by the therapist
  Arms: Group A (Hydrodilation+Spencer Technique )
Procedure: Passive Stretching — The low intensity stretches will be given in supine for all the movements ie Flexion ,Abduction , Internal Rotation and External Rotation for 5 repititions with 30 sec hold.
  Arms: Group B (Hydro dilation+ Passive Stretching)

SUMMARY:
Adhesive Capsulitis is a common Musculoskeletal disorder characterized by pain and progressive joint restriction in capsular pattern. Adhesive capsulitis can be managed by both conservative and non conservative treatment. The Spencer technique and hydrodilation are two treatment approaches used to restore range of motion in adhesive capsulitis.

The Spencer technique is a form of physical therapy that involves joint mobilizations and manual stretching exercises. It aims to improve shoulder mobility and reduce pain by addressing the tightness and stiffness in the shoulder capsule and surrounding tissues.

Hydrodilation, on the other hand, is a procedure where a saline solution is injected into the shoulder joint to distend the capsule. This distention helps stretch the tight tissues and break up adhesions, facilitating improved range of motion.

DETAILED DESCRIPTION:
Adhesive capsulitis, also subsequently known as Frozen shoulder is a musculoskeletal disorder characterized by painful and progressive joint restriction in capsular pattern. It has a prevalence of 2 to 5% in general population and the incidence is more in females mostly aged 40 to 60 years mostly suffering from Diabetes Mellitus. Adhesive Capsulitis can be classified into three phases; Freezing (painful), Frozen (stiffening) and Thawing (resolution phase). The treatment protocol is planned such to improve the range of motion and reduce pain. Various treatment regimes are followed for treatment of adhesive capsulitis, either it be in medical field, physical therapy or in worst cases surgical treatments too.

Hydrodilation, a medical procedure which involves injecting a fluid (mainly normal saline) into the joint space which expands the space breaking up scar tissue and loosening the joint. This method is being widely used in isolation or in combination with other methods to treat Adhesive capsulitis.

Spencer technique on another hand is a physical therapy technique which in isolation or in conjunction with other treatments is used to treat patients with adhesive capsulitis. Spencer muscle energy technique is a seven 7 step procedure which consists of shoulder extension with elbow flexed, shoulder flexion with elbow flexed, circumduction with compression, circumduction with traction, Abduction then adduction with external rotation and glenohumeral pump.

Hence the current study will investigate the effects of Spencer technique following hydrodilation in patients with Adhesive Capsulitis.

The study includes subjects with unilateral adhesive capsulitis, 40-60 years of age both male and female and have undergone Hydrodilation. The selction of subjects will be using non probability purposive sampling technique. Participants will be randomized using sealed envelope method and allocated to one of two groups.

The data collection tool for pain is VAS, for ROM is Goniometer and for disability is SPADI.

The time duration for treatment protocol is total of 12 sessions, 3 sessions per week. Exercise is done 3 to 5 times with rest periods.

ELIGIBILITY:
Inclusion Criteria:

* Patients with diagnosed unilateral Adhesive Capsulitis and have undergone Hydrodilation. --Includes both genders
* Age 40 to 60 years. Exclusion Criteria
* Population who have recently undergone major shoulder injury or surgery, had fracture or open wound or there is reduction of Glen humeral ROM due to any other cause other than Adhesive Capsulitis

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-07-20 (Actual); Primary Completion 2024-10-01 (Actual); Study Completion 2024-10-31 (Estimated)

PRIMARY OUTCOMES:
Shoulder ROM | 4 weeks
  Range of Motion will be measured using the universal Goniometer which is 0 to 180 degree for half circle model or 0 to 360 degree for full circle models.
Pain Intensity | 04 Weeks
  Pain will be assessed using Visual Analog scale which is 0-100 item scale.

SECONDARY OUTCOMES:
Shoulder Disability | 4 weeks
  Shoulder Disability will be assessed using shoulder pain and disability index.

CONTACTS AND LOCATIONS:
Locations (1):
- Foundation University College of Physical Therapy, Rawalpindi, Punjab Province, Pakistan